CLINICAL TRIAL: NCT01870830
Title: Nocturnal Breathing and Sleep in Patients With Chronic Obstructive Pulmonary Disease Staying at Altitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2013-088B
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A: low-intermediate-high altitude (Other): Altitude exposure sequence A, 490-1650-2590m
  Interventions: Other: Altitude exposure
- B: low-high-intermediate altitude (Other): Altitude exposure sequence B, 490-2590-1650m
  Interventions: Other: Altitude exposure
- C: intermediate-high-low altitude (Other): Altitude exposure sequence C, 1650-2590-490m
  Interventions: Other: Altitude exposure
- D: high-intermediate-low altitude (Other): Altitude exposure sequence D, 2590-1650-490m
  Interventions: Other: Altitude exposure

INTERVENTIONS:
Other: Altitude exposure — Stay at different altitudes: 490, 1650, 2590 m

SUMMARY:
The purpose of this study is to evaluate whether nocturnal breathing and sleep of patients with chronic obstructive pulmonary disease (COPD) are disturbed during a stay at moderate altitude.

DETAILED DESCRIPTION:
This randomized cross-over trial evaluates the hypothesis that patients with chronic obstructive pulmonary disease experience nocturnal hypoxemia, periodic breathing and sleep disturbances when staying at moderate altitude. Sleep studies and clinical evaluations will be performed during 2 days in Zurich (490 m, low altitude baseline) and during 2 days at Davos Clavadel (1650 m), and 2 days at Davos Jakobshorn (2590 m).

ELIGIBILITY:
Inclusion Criteria:

* chronic obstructive pulmonary disease (COPD), GOLD grade 2-3
* residents at low altitude (<800 m)

Exclusion Criteria:

* Unstable condition, COPD exacerbation
* Mild (GOLD 1) or very severe COPD (GOLD 4)
* requirement for oxygen therapy at low altitude residence
* hypoventilation
* pulmonary hypertension
* more than mild or unstable cardiovascular disease
* use of drugs that affect respiratory center drive
* internal, neurologic or psychiatric disease that interfere with protocol compliance including current heavy smoking (>20 cigarettes per day), inability to perform 6 min walk test.
* previous intolerance to moderate altitude (<2600m).
* Exposure to altitudes >1500m for >2 days within the last 4 weeks before the study.
* Pregnant or nursing patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in mean nocturnal oxygen saturation from baseline measured at 490 m | Change in mean nocturnal oxygen saturation from 490 m baseline during 2 days at 2590 m
  mean nocturnal oxygen saturation measured by pulse oximetry
Change in apnea/hypopnea index from baseline measured at 490 m | Change in apnea/hypopnea index from 490 m baseline during 2 days at 2590 m
  apnea/hypopnea index measured by polysomnography

SECONDARY OUTCOMES:
Change in mean nocturnal oxygen saturation from baseline measured at 490 m | Change in mean nocturnal oxygen saturation from 490 m baseline during 2 days at 1650 m
  apnea/hypopnea measured by polysomnography
Change in apnea/hypopnea index from baseline measured at 490 m | Change in apnea/hypopnea index from 490 m baseline during stay at 1650 m
  apnea/hypopnea index measured by polysomnography
Change in subjective sleep quality from baseline measured at 490 m | Change in subjective sleep quality from 490 m during 2 days at 2590 m
  Visual analog scale of sleep quality
Change in subjective sleep quality from baseline measured at 490 m | Change in subjective sleep quality from 490 m baseline during 2 days at 1650 m
  Visual analog scale of sleep quality
Change in reaction time from baseline measured at 490 m | Change in reaction time from 490 m baseline during 2 days at 2590 m
  psychomotor vigilance test reaction time
Change in reaction time from baseline measured at 490 m | Change in reaction time from 490 m baseline during 2 days at 1650 m
  Psychomotor vigilance test reaction time

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Chair — University Hsopital Zurich, Switzerland; Tsogyal D Latshang, MD, Principal Investigator — University Hospital, Zürich
Locations (1):
- University Hospital Zurich, Pulmonary Division, Zurich, Switzerland

REFERENCES:
- [Derived] Latshang TD, Tardent RPM, Furian M, Flueck D, Segitz SD, Mueller-Mottet S, Kohler M, Ulrich S, Bloch KE. Sleep and breathing disturbances in patients with chronic obstructive pulmonary disease traveling to altitude: a randomized trial. Sleep. 2019 Jan 1;42(1). doi: 10.1093/sleep/zsy203. PMID 30517695